CLINICAL TRIAL: NCT04754256
Title: Causes of Appetite Loss in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Type: Observational
Sponsor: Jens Rikardt Andersen (Other)
Responsible Party: Sponsor-Investigator, Jens Rikardt Andersen, Lecturer, University of Copenhagen
Organization: University of Copenhagen (Other)
Other Study IDs: H-20054785
Record Dates: First submitted 2021-02-09; First posted 2021-02-15 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Council of Nutrition Appetite Questionnaire - test for applicability in Danish COPD patients — Council of Nutrition Appetite Questionnaire - test for applicability in Danish COPD patients and for correlation of scores with lung function, CAT-score and other

SUMMARY:
The project looks at causes of appetite loss in patients with COPD. It is know that active systemic inflammation can lead to appetite loss and COPD is classified as a disease lead by inflammation. But it has never been investigated if the patient with COPD has other causes of appetite loss such as physical, psychological or social barriers for not reaching a sufficient dietary intake.

The study uses a homemade questionnaire, the CAT-scale and the CNAQ-score to evaluate the extent of appetite loss and certain demographic characteristics of the participants. There will be made correlation analysis for CNAQ-score and continuous variables and there will be tested for significant differences between the group who scores as low appetite and the group that scores with a normal appetite via CNAQ.

The second part of the study invites patients to participate in a semi-structured interview, that focuses on the patient's experience with appetite loss, meals and food. The interviews will be transcribed and analysed.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: COPD patients found in Danish Facebook support group
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
CNAQ-score | 6 months
  Appetite questionnaire to divide participants in either normal appetite or loss of appetite

CONTACTS AND LOCATIONS:
Locations (1):
- University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided